CLINICAL TRIAL: NCT03252041
Title: MRI & MRV in Pelvic Congestion Syndrome in Females
Acronym: PCS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed AbuDeif Sayed, Dr, Assiut University
Other Study IDs: MRI & MRV in PCS
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Pelvic Pain Syndrome
Keywords: PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — Magnetic Resonance imaging modalities and sequences in pelvic congestion syndrome

SUMMARY:
To investigate the feasibility of MRI and MRV in diagnosis of pelvic congestion syndrome.

DETAILED DESCRIPTION:
In the past, a diagnosis of chronic pelvic pain left many women frustrated with few treatment options and a lack of available resources. Their physicians were likewise perplexed, despite the endless acquisition of negative laboratory and imaging data as well as inconclusive consultations obtained. In the last 10 years, improved scientiﬁc understanding and increased physician awareness have lessened the confusion surrounding this condition and its distinct association with pelvic congestion syndrome (PCS). Furthermore, reﬁnements of medical and minimally invasive surgical solutions give affected patients more therapeutic choices today.

Since anatomical venous variations in the pelvis are common, it is important to know the anatomy of these vessels for treatment planning. Imaging is critical in the evaluation of pelvic varices, both to differentiate them from other condition and also because pelvic varices may be secondary to serious underlying pathology, such as inferior vena caval obstruction, portal hypertension, increased pelvic blood flow, and vascular malformations.

The diagnosis of PCS has usually been suggested by duplex ultrasound (US), but ultrasound imaging does not readily show the gonadal veins. Phlebography is the "gold standard" for anatomic diagnostic studies. Related mortality and morbidity are low, but patient discomfort and costs make this an unattractive routine method of diagnosis. Magnetic resonance imaging (MRI) can usually demonstrate pelvic and ovarian varices, as well as the gonadal veins.

In this prospective study, we will investigate the feasibility of using magnetic resonance venography (MRV) in the diagnosis of PCS and evaluated its accuracy and reliability in comparison to phlebography.

ELIGIBILITY:
Inclusion Criteria:

* All patients with signs and symptoms of PCS.

Exclusion Criteria:

* Patients with general contraindications to MRI as presence of any para-magnetic substance as pacemakers, or in severely ill patients or those with claustrophobia, arrhythmic patients.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — In the past, a diagnosis of chronic pelvic pain left many women frustrated with few treatment options and a lack of available resources. Their physicians were likewise perplexed, despite the endless acquisition of negative laboratory and imaging data as well as inconclusive consultations obtained. In the last 10 years, improved scientiﬁc understanding and increased physician awareness have lessened the confusion surrounding this condition and its distinct association with pelvic congestion syndrome (PCS). Furthermore, reﬁnements of medical and minimally invasive surgical solutions give affected patients more therapeutic choices today.
Study Population: females with chronic lower abdominal pain, signs and symptoms of pelvic congestion syndrome
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
MRI and MRV in pelvic congestion syndrome in females. | one year
  To investigate the feasibility of MRI and MRV in diagnosis of pelvic congestion syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Galal, ass prof, Study Chair — Assiut University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
to be shared when finished